CLINICAL TRIAL: NCT06152367
Title: Phase I/II Trial In Stage III/IV Malignant Melanoma Using Autologous Dendritic Cells Loaded With Tumor Cell Lysates And Low Doses Of Proleukin
Brief Title: Immunization With Autologous Dendritic Cells and Tumor Lysates in Melanoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCHD04T2026
Record Dates: First submitted 2023-09-27; First posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Stage III Malignant Melanoma of Skin AJCC V6; Stage IV Malignant Melanoma of Skin
MeSH Terms: conditions — Melanoma | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAPCells (Experimental): Patients are immunized with four doses of TAPCells (20x106), days 0, 10, 20, and 50 complemented with low doses 2·4×106 IU/m2 rhIL-2 (Proleukin®) (Chiron Emeryville, CA, USA), injected s.c. days 2, 3, and 4 after a second, third, and fourth vaccination.
  Interventions: Biological: TAPCells vaccine

INTERVENTIONS:
Biological: TAPCells vaccine — Patients are immunized with four doses of TAPCells (20x106), days 0, 10, 20, and 50 complemented with low doses 2·4×106 IU/m2 rhIL-2 (Proleukin®) (Chiron Emeryville, CA, USA), injected s.c. days 2, 3, and 4 after a second, third, and fourth vaccination.
  Other Names: Proleukin

SUMMARY:
Implementing this protocol has its ethical justification in that patients with metastatic melanoma, once tumor invasion has reached beyond the lymph node barrier, cannot possibly be treated satisfactorily with traditional surgery methods, radiotherapy, or conventional available chemotherapy. The disseminated tumor is refractory to all standard treatments. Almost 100% of patients who develop distant metastases will die from their disease, either from complications or cachexia. Therefore, immunotherapy based on immunological stimulation with immunocompetent dendritic cells, added to immunological reinforcement with IL-2, can, according to the evidence emanating from ongoing clinical protocols, produce a prolongation of survival with better quality and, in some cases, with partial or total regression of the tumor.

General objective: It is to study the clinical and immunological response of patients treated with vaccines based on autologous dendritic cells loaded with tumor antigens, derived from allogeneic melanoma extracts, in combination or not, with intercalated low doses of recombinant human interleukin 2 (rhIL2) PROLEUKIN ® (aldesleukin). MAIN SPECIFIC OBJECTIVE: - SAFETY: Safety in administering dendritic cell preparation; local and systemic toxicity estimation. Determination of adverse reactions such as fever, nausea, allergy, neurological and cardiovascular symptoms. Local toxicity in the administration area. - MEASUREMENT OF THE IMMUNE RESPONSE: Based on in vivo and in vitro parameters: - In vivo response: Measure the type IV Delayed Hypersensitivity (DTH) response. It consists of a crossover test in which the response is compared to tissue interaction in vivo between dendritic cells sensitized with tumor extracts and their respective control unloaded dendritic cells. - In vitro response: ELISPOT assays, measurement of IFN-γ gamma production in peripheral blood of treated patients. Compare the specific immune response after each cycle of therapy through measurement of IFN-γ production by tumor-specific CTL. Cytotoxic radioactive chromium release assays to measure anti-tumor response mediated by CTL and NK. ELISA assays for quantifying cytokines (IFN-γ, IL-10) in patient serum after each cycle of therapy.

DETAILED DESCRIPTION:
Vaccination of Melanoma Patients Using DCs Loaded with Allogeneic Melanoma Extracts.

In Chile, this study constitutes the first phase I clinical trial for treating advanced malignant melanoma using dendritic cell vaccines loaded with allogeneic tumor extracts complemented or not with low doses of rIL-2. Since chemotherapy and radiotherapy only offer palliative effects in advanced melanoma, resulting in an inferior prognosis for these patients, the trial intends to develop a protocol that would adapt to the reality of Chile, allowing for a combination of high technology and low costs.

After obtaining approval from the human research ethics committee from Universidad de Chile, 86 patients will be recruited who will be duly informed about the scope of these protocols and the realistic prospects of success. The participants then will undergo a comprehensive health check to assess their overall health. The participants will undergo a leukapheresis at the blood bank of the Clinical Hospital of the University de Chile. Peripheral blood mononuclear cells (PBMCs) will be separated using a Ficoll-Hypaque gradient in the laboratory of Antitumor Immunology at the Institute of Biomedical Sciences, Faculty of Medicine of the University de Chile. Some of the cells will be cryopreserved in liquid nitrogen for future use. Approximately 1.8x108 PBMCs will be placed in 6-well culture plates and incubated at 37°C and 7% CO2 for two hours. The suspended cells, peripheral blood lymphocytes (PBLs), will be removed and frozen for later use. The monocytes adhering to the plastic will be incubated for seven days in a serum-free culture medium (AIM-V therapeutic, GIBCO, BRL) in the presence of 500 U/ml of IL-4 and 800 U/ml of GM-CSF. On the sixth day, the DCs will be pulsed with tumor extracts from allogeneic melanoma cell lines, previously checked for sterility, and incubated for 6 hours at 37°C and 7% CO2, followed by maturation stimulus with TNF-alpha for 12 to 18 hours. Mature DCs will be characterized by flow cytometry. Approximately 10 to 20 x 106 pulsed DCs will be subcutaneously injected. This routine will be repeated weekly for at least four times and a maximum of 6 times. After the fourth dose, the participant's general condition, possible clinical regressions, adverse side effects, and the effects of the treatment on the immune system will be evaluated. This evaluation will be done through in vivo delayed-type hypersensitivity (DTH) assays using melanoma extracts and their respective controls. Planned in vitro assays for immune response measuring will include the detection of anti-melanoma CTL precursors by ELISPOT, cytokine production, proliferation assays, and quantifying the CD4/CD8 ratio by flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed melanoma of the skin: Breslow, Clark, histological type. Location of the primary, clinical, or pathological regional status.
* Complete staging demonstrating the presence of distant metastases, either visceral or in soft tissues or bone tissue: Brain, Lung, Abdomen, and Pelvis CT and bone scintigraphy.
* Objectively measurable disease by clinical or radiological means
* Karnofsky's Performance Status is more significant than 70%
* Life expectancy greater than three months
* Patients over 18 years old
* Informed consent from the patient to participate in the protocol

Exclusion Criteria:

* Age greater than or equal to 65 years
* Ongoing active infections, including viral immunodeficiency
* Previous chemotherapy within less than two months
* Concomitant malignant tumors (e.g., Chronic Lymphocytic Leukemia, etc.)
* Uncontrolled concomitant diseases (Hypertension, unstable Diabetes mellitus, renal diseases requiring dialysis)
* Situations or conditions requiring urgent surgical intervention, such as intestinal obstruction due to metastasis
* Pregnancy or lactation
* Concurrent participation in other therapeutic research protocols
* Any condition that compromises the objectives of this study.

Removal Criteria from the Study:

* By the patient's decision to discontinue the study.
* Intolerable adverse reactions, according to WHO Criteria Grading Toxicities
* Intercurrent illness that may compromise the patient's life or interfere with the treatment study evaluation
* Requirements for concomitant medication that may interfere with study results.
* Failure to complete the study entirely
* Failure to follow up on the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2001-01-30 (Actual); Primary Completion 2004-10-09 (Actual); Study Completion 2004-10-09 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events [safety and tolerability] | Every four weeks the first year after treatment. Every two months during the second year after treatment.
  Safety in administering dendritic cell preparations; Toxicity will be evaluated during every immunization and DTH test, using the NCI Common Terminology Criteria for Adverse Events Cancer Therapy Evaluation Program (CTCAE, Bethesda, MD, USA) v.3.0. In addition, patients will have a 24-h emergency phone number to report adverse events. Local and systemic toxicity estimation will be evaluated.
Local immune response measurement by DTH | Every four weeks the first year after treatment. Every two months during the second year after treatment.
  Measuring the Delayed-Type Hypersensitivity response (DTH). It involves a cross-test comparing in vivo tissue response after injecting sc. tumor cell lysates used in the vaccine, PBS, or positive control antigenic mix. The test will be performed before the treatment and 30 days after the fourth dose. A positive DTH reaction is defined as skin erythema or induration ≥ 5 mm 48 hours after injection.
Systemic immune response measurement in PBMC | Every four weeks the first year after treatment. Every two months during the second year after treatment.
  Measuring of multiple cytokine release (IFN-γ, IL-17, TGF-b, IL-10, and TNF-a) in patient PBMC subpopulations by flow cytometry analysis. Statistically significant increases in IFN-g and IL-17 will be considered positive immune responses. Increases in TGF-b, IL-10, and TNF-a will be considered tolerogenic responses. PBMC subpopulation analysis will be performed after in vitro re-stimulations.
Systemic IFN-γ response measurement in serum | Every four weeks the first year after treatment. Every two months during the second year after treatment.
  Measuring of IFN-γ release in patient serum by ELISA assay. Statistically significant increases in IFN-g serum levels will be considered positive immune responses.
Systemic IL-17 response measurement in serum | Every four weeks the first year after treatment. Every two months during the second year after treatment.
  Measuring of IL-17 release in patient serum by ELISA assay. Statistically significant increases in IL-17 serum levels will be considered positive immune responses.
Systemic TGF-b response measurement in serum | Every four weeks the first year after treatment. Every two months during the second year after treatment.
  Measuring of TGF-b release in patient serum by ELISA assay. Statistically significant increases in TGF-b serum levels will be considered tolerogenic immune responses.
Systemic IL-10 response measurement in serum | Every four weeks the first year after treatment. Every two months during the second year after treatment.
  Measuring of IL-10 release in patient serum by ELISA assay. Statistically significant increases in IL-10 serum levels will be considered tolerogenic immune responses.
Systemic TNF-a response measurement in serum | Every four weeks the first year after treatment. Every two months during the second year after treatment.
  Measuring of TNF-a release in patient serum by ELISA assay. Statistically significant increases in TNF-a serum levels will be considered tolerogenic immune responses.
Systemic cytotoxic T cell-mediated tumor-specific IFN-g release | Every four weeks the first year after treatment. Every two months during the second year after treatment.
  Measuring IFN-g production by tumor antigen in vitro-activated tumor-specific CTLs derived from peripheral blood of treated patients after each vaccine injection by IFN-g ELISPOT assays.
Systemic cytotoxic T cell-mediated anti-tumor cell cytotoxicity | Every four weeks the first year after treatment. Every two months during the second year after treatment.
  Measuring cytotoxicity by tumor antigen in vitro activated tumor-specific CTLs derived from peripheral blood of treated patients after each vaccine injection by radioactive chromium releases cytotoxic assays.

SECONDARY OUTCOMES:
Overall survival | Every four weeks the first year after treatment. Every two months during the second year after treatment.
  Post-vaccination OS will be defined as the mean time that patients are still alive after the first vaccine dose injection using Kaplan-Meier survival analysis.
Progression-free survival | Every four weeks the first year after treatment. Every two months during the second year after treatment.
  PFS is defined as the meantime that a patient showed stable disease after first vaccine dose.Time from treatment until disease recurrence (or death) using Kaplan-Meier survival analysis.
Clinical response measurement | Every four weeks the first year after treatment. Every two months during the second year after treatment.
  To observe the objective response rate. Patients were defined as immunologic responders if they displayed activity against TRIMEL in DTH assays. Stable disease (SD) will be defined as less than 25% change in tumor size and absence of new lesions during a 6-week period. Inversely, progressive disease (PD) will be defined as more than 25% increase in the perpendicular diameter of any measurable tumor, appearance of new lesions by imaging examination, and/or worsening of general condition.
Global health status scores measurement | Evaluated at immunization 1 (day 0; baseline level), 3 (day 20) and 4 (day 50), and also at DTH test (day 80)
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) is a 30-item questionnaire, validated in Chile in Spanish language, that will completed by the patients. It include both multi-item scales and single-item measures. It include five functional scales, three symptom scales, six single items, and a Global Health Status/Quality of Life (GHS/QoL) scale.
  The GHS/QoL scale has seven possible response scores ranging from 1 (very poor) to 7 (excellent), which will be averaged and transformed to a 0-100 scale. A higher score on this scale indicated a better quality of life.
  The change from baseline in GHS/QoL scores will be calculated. A positive change from baseline indicated improvement in the patient's quality of life.
Physical functioning scale scores measurement | Evaluated at immunization 1 (day 0; baseline level), 3 (day 20) and 4 (day 50), and also at DTH test (day 80)
  The EORTC QLQ-C30 pain symptom scale is one of the symptom scales in the questionnaire, which measured the severity of pain experienced by the patient. The pain symptom scale consist in two items, one measuring the severity of pain and the other measuring the use of painkillers. The items will be rated on a 4-point scale ranging from 1="not at all" to 4="very much". The scores for each item will be summed and transformed to a 0 to 100 scale (higher scores indicating more severe pain).
  The change from baseline in pain symptom scale scores will be calculated. A negative change from baseline indicated improvement.
Pain symptom scale scores measurement | Evaluated at immunization 1 (day 0; baseline level), 3 (day 20) and 4 (day 50), and also at DTH test (day 80)
  The EORTC QLQ-C30 physical functioning scale measures a patient's ability to carry out daily activities and tasks requiring physical exertion. It consist in five questions asking patients to rate their level of physical functioning, with response options ranging from 1="not at all" to 4="very much". The scores for each item will summed and transformed to a 0 to 100 scale, with higher scores indicating better physical functioning.
  The change from baseline in physical functioning scale scores will be calculated. A positive change from baseline indicated improvement in physical functioning.The GHS/QoL scale has seven possible response scores ranging from 1 (very poor) to 7 (excellent), which will be averaged and transformed to a 0-100 scale. A higher score on this scale indicated a better quality of life.
  The change from baseline in GHS/QoL scores will be calculated. A positive change from baseline indicated improvement in the patient's quality of life.
Performance status response | Every four weeks the first year after treatment. Every two months during the second year after treatment.
  Percentage of patients with a 20% or more significant increase in activity measured by the Karnofsky index

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Salazar-Onfray, PhD, Principal Investigator — FACULTY OF MEDICINE, Universidad de Chile
Locations (1):
- Faculty of Medicine, University of Chile, Santiago, RM, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aguilera R, Saffie C, Tittarelli A, Gonzalez FE, Ramirez M, Reyes D, Pereda C, Hevia D, Garcia T, Salazar L, Ferreira A, Hermoso M, Mendoza-Naranjo A, Ferrada C, Garrido P, Lopez MN, Salazar-Onfray F. Heat-shock induction of tumor-derived danger signals mediates rapid monocyte differentiation into clinically effective dendritic cells. Clin Cancer Res. 2011 Apr 15;17(8):2474-83. doi: 10.1158/1078-0432.CCR-10-2384. Epub 2011 Feb 3. PMID 21292818
- [Background] Duran-Aniotz C, Segal G, Salazar L, Pereda C, Falcon C, Tempio F, Aguilera R, Gonzalez R, Perez C, Tittarelli A, Catalan D, Nervi B, Larrondo M, Salazar-Onfray F, Lopez MN. The immunological response and post-treatment survival of DC-vaccinated melanoma patients are associated with increased Th1/Th17 and reduced Th3 cytokine responses. Cancer Immunol Immunother. 2013 Apr;62(4):761-72. doi: 10.1007/s00262-012-1377-3. Epub 2012 Dec 15. PMID 23242374
- [Background] Tittarelli A, Gonzalez FE, Pereda C, Mora G, Munoz L, Saffie C, Garcia T, Diaz D, Falcon C, Hermoso M, Lopez MN, Salazar-Onfray F. Toll-like receptor 4 gene polymorphism influences dendritic cell in vitro function and clinical outcomes in vaccinated melanoma patients. Cancer Immunol Immunother. 2012 Nov;61(11):2067-77. doi: 10.1007/s00262-012-1268-7. Epub 2012 May 3. PMID 22552381
- [Background] Garcia-Salum T, Villablanca A, Matthaus F, Tittarelli A, Baeza M, Pereda C, Gleisner MA, Gonzalez FE, Lopez MN, Hoheisel JD, Norgauer J, Gebicke-Haerter PJ, Salazar-Onfray F. Molecular signatures associated with tumor-specific immune response in melanoma patients treated with dendritic cell-based immunotherapy. Oncotarget. 2018 Mar 30;9(24):17014-17027. doi: 10.18632/oncotarget.24795. eCollection 2018 Mar 30. PMID 29682201
- [Result] Lopez MN, Pereda C, Segal G, Munoz L, Aguilera R, Gonzalez FE, Escobar A, Ginesta A, Reyes D, Gonzalez R, Mendoza-Naranjo A, Larrondo M, Compan A, Ferrada C, Salazar-Onfray F. Prolonged survival of dendritic cell-vaccinated melanoma patients correlates with tumor-specific delayed type IV hypersensitivity response and reduction of tumor growth factor beta-expressing T cells. J Clin Oncol. 2009 Feb 20;27(6):945-52. doi: 10.1200/JCO.2008.18.0794. Epub 2009 Jan 12. PMID 19139436

DOCUMENTS (2):
  • Study Protocol (2001-07-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT06152367/Prot_000.pdf
  • Informed Consent Form (2001-04-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT06152367/ICF_001.pdf